CLINICAL TRIAL: NCT03072823
Title: Omega-3 Polyunsaturated Fatty Acids on Major Depressive Disorder in Patients With Cardiovascular Diseases: a Double-blind Placebo-controlled Therapeutic Trial
Brief Title: Omega-3 Polyunsaturated Fatty Acids on Major Depressive Disorder in Patients With Cardiovascular Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Pei-Chen Chang, Attending Physician, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH104-REC2-059
Record Dates: First submitted 2017-02-24; First posted 2017-03-07 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Cardiovascular Diseases; Major Depressive Disorder
Keywords: CVDs; cardiovascular diseases; n-3 polyunsaturated fatty acids; depression
MeSH Terms: conditions — Cardiovascular Diseases; Depressive Disorder, Major; Depression | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- n-3 polyunsaturated fatty acids (Active Comparator): n-3 polyunsaturated fatty acids dosage of 2 g of Eicosapentaenoic acid(EPA) and 1 g of Docosahexaenoic acid (DHA).
  Interventions: Dietary Supplement: n-3 Polyunsaturated fatty acid
- placebo (Placebo Comparator): olive oil ethyl esters
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: n-3 Polyunsaturated fatty acid — 2 g of Eicosapentaenoic acid (EPA) and 1 g of Docosahexaenoic acid (DHA)
  Arms: n-3 polyunsaturated fatty acids
Dietary Supplement: placebo — olive oil ethyl esters
  Arms: placebo

SUMMARY:
N-3 polyunsaturated fatty acids(N-3 PUFAs) is important in balancing the immune function and physical health by reducing membrane arachidonic acid (AA) and prostaglandin E2 (PGE2) synthesis, which might be linked to the somatic manifestations physical morbidity, such as Cardiovascular disease in depression. n-3 polyunsaturated fatty acids appears to be a promising treatment that is safe, beneficial to patients with Cardiovascular disease and depression. In this proposal, investigators aim the test the hypothesis that n-3 polyunsaturated fatty acids will be more effective than placebo in treating Cardiovascular disease patients with major depression after 12 weeks of intervention.

DETAILED DESCRIPTION:
This is a 3-year study and a randomized, double-blind, and placebo controlled Clinical the study. investigators plan to enroll 60 subjects from cardiovascular department of China Medical University Hospital.Participants will be randomized into omega-3 polyunsaturated fatty acids or placebo group.The intervention period is 12 weeks. Evaluation of the depressive symptoms ( using Hamilton Depression Scale, HAM-D, and Beck Depression Inventory, BDI ) of the subjects who are enrolled into the study will take place at -1st, 0, 2nd, 4th, 8th, 12th week. The plasma level of n-3 polyunsaturated fatty acids, chemokines/cytokines, and Electrocardiogram will also be measured at the beginning and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Cardiovascular disease patients
2. The Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for major depressive disorder.
3. Capacity and willingness to give written informed consent.

Exclusion Criteria:

1. cognitive impairment (Mini-mental state examination score <24)
2. comorbid psychiatric disorders, psychosis, high risk of suicide, current substance use
3. an acute coronary syndrome within previous 2 months, left ventricular ejection fraction (LVEF)<30%, advanced malignancy, or physical inability to participate
4. use of antidepressants, anticonvulsants, lithium, or n-3 polyunsaturated fatty acids supplements
5. coagulation disorders or sensitivity to n-3 polyunsaturated fatty acids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Scale(HAM-D) score at 3 months | Week 0, Week 2, Week 4 Week 8, Week 12
Change in Beck's Depression Inventory(BDI) score at 3 months | Week 0, Week 2, Week 4 Week 8, Week 12

SECONDARY OUTCOMES:
Electrocardiogram (EKG) | Week 0, Week 2, Week 4 Week 8, Week 12
mini nutritional assessment (MNA) score | Week 0, Week 2, Week 4 Week 8, Week 12
Adverse effects | Week 0, Week 2, Week 4 Week 8, Week 12
plasma level of n-3 polyunsaturated fatty acids | Week 0, Week 12
plasma cytokine/chemokine | Week 0, Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taiwan

REFERENCES:
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851